CLINICAL TRIAL: NCT01168557
Title: Stress Echo and Electric Impedance Tomography (EIT) Pilot Study to Investigate the Influence of Cardiac Output on Parameters of the EIT
Brief Title: Stress Echo and Electric Impedance Tomography (EIT) Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Stress Echo - EIT
Record Dates: First submitted 2010-07-22; First posted 2010-07-23 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Electric Impedance Tomography; Stress Echocardiography; Cardiac Output; Ventilation; Perfusion
Keywords: electric impedance tomography; stress-echocardiography; ventilation; perfusion
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stress-Echo and EIT (Experimental): Patients who routinely undergo stress-echocardiography will additionally be measured by EIT using a rubber belt, which will be placed around their chest
  Interventions: Device: EIT (Electrical Impedance Tomography)

INTERVENTIONS:
Device: EIT (Electrical Impedance Tomography) — EIT measurement; concomitant to stress echocardiography (about 45 minutes) EIT measurements (1 minute) are performed at rest, at low dobutamine stress, at peak and at relaxation

SUMMARY:
Electric Impedance Tomography (EIT) is a technique based on the injection of small currents and voltage measurements using electrodes on the skin surface generating cross-sectional images representing impedance change in a slice of the thorax.It is a radiation free, non- invasive and portable lung imaging technique. Impedance changes in lung ventilation as well as in lung perfusion can be shown. To investigate lung perfusion by EIT measurements, cardiac output measured by routinely undergone stress echocardiography at rest and stress are compared to parameters measured by EIT.

DETAILED DESCRIPTION:
In 15 patients who routinely have to undergo stress echocardiography Electric Impedance Tomography (EIT) measurements are performed parallel to measurements of cardiac output at rest, low stress generated by a dosage of 10µg dobutamine, at peak generated by a dosage between 20-40µg dobutamine (individually)and at relaxation(pulse <100). Therefore prior to the examination a rubber belt with 16 integrated electrocardiographic electrodes is placed around the thorax at the fifth or sixth intercostal space, connected with an EIT device. EIT data are generated by application of a small alternating electrical current of 5mA and 50kHz and are stored and analyzed offline on a personal computer. Changes due to ventilation as well as changes due to perfusion will be measured by EIT. Cardiac output will be retrospectively compared to parameters of the EIT. EIT data are stored in a database and pseudonymized evaluated in relationship to routinely measured stress echocardiography data.

ELIGIBILITY:
Inclusion Criteria:

* male patients >18 years who routinely have to undergo stress echocardiography
* ejection fraction >50%
* able to give informed consent

Exclusion Criteria:

* restrictive lung diseases
* active implants and heart pace makers and implanted converter defibrillator
* foreign metallic objects in the thorax
* Not adequate quality of imaging of stress echocardiography

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2010-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
influence of cardiac output on EIT measurements (feasibility) | single measurement of 45 minutes
  It will be investigated if a change in cardiac output, which is measured by stress-echocardiography by dobutamine, has an influence on the parameters determined by EIT measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Krueger, MD, Assoc. Prof., Principal Investigator — RWTH Aachen University of Cardiology, Pneumology and Angiology, Aachen, NRW, Germany
Locations (1):
- Medical Clinic I, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany